CLINICAL TRIAL: NCT02971475
Title: Extracorporeal Shock Wave Lithotripsy Versus Extracorporeal Shock Wave Lithotripsy Combined With Endoscopic Treatment for Painful Calcified Chronic Pancreatitis
Brief Title: ESWL Versus ESWL and Endoscopic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Deputy Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160801
Record Dates: First submitted 2016-09-05; First posted 2016-11-23 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Pancreatitis
Keywords: Extracorporeal Shock Wave lithotripsy(ESWL); Endoscopic Retrograde Cholangiopancreatography(ERCP); chronic pancreatitis; pain relief
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic | interventions — Lithotripsy; Cholangiopancreatography, Endoscopic Retrograde; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESWL alone (Experimental): Patients in this group would be treated with extracorporeal shock wave lithotripsy only. Otherwise, extra endoscopic procedures will be carried out in case of continuous and aggravated pain. Analgesics will be administrated as needed and recorded.
  Interventions: Procedure: extracorporeal shock wave lithotripsy; Drug: Analgesics
- ESWL combined with ERCP (Active Comparator): People in this group would be treated with ESWL followed be endoscopic drainage of the main pancreatic duct in 48 hours. Analgesics will be administrated as needed and recorded.
  Interventions: Procedure: endoscopic drainage of the main pancreatic duct; Drug: Analgesics

INTERVENTIONS:
Procedure: extracorporeal shock wave lithotripsy — People in this group would be treated with ESWL only.
  Other Names: ESWL
  Arms: ESWL alone
Procedure: endoscopic drainage of the main pancreatic duct — People in this group would be treated with ESWL followed be endoscopic drainage in 48 hours.
  Other Names: ERCP
  Arms: ESWL combined with ERCP
Drug: Analgesics — Analgesics administrated include morphine, buprenorphine, pethidine, tramaldol, metamizole and acetylsalicylacid. They will only be administrated as needed.

SUMMARY:
The study wants to compare ESWL alone with ESWL and endoscopic drainage of the MPD for treatment of pain in chronic pancreatitis.

DETAILED DESCRIPTION:
The combination mode of ESWL and ERCP is an established method of treatment of painful obstructive calcified chronic pancreatitis. However, the investigators notice that patients after ESWL alone in calcified CP is followed by spontaneous elimination of stone fragments and pain relief. Inui reported that 40% of 555 patients spontaneous eliminate stone fragments. Dumonceau found that combining systematic endoscopy with ESWL adds to the cost of patient care, without improving the outcome of the pancreatic pain.

So the investigators design such a prospective and randomized controlled trial. People diagnosed with uncomplicated painful chronic pancreatitis and calcifications obstructing the MPD will be randomly assigned to the ESWL or endoscopy group according to a table of random numbers.

ESWL will be performed in all patients using a electromagnetic lithotriptor. ESWL sessions will be repeated if necessary, until stone fragmentation is obtained. Patients in the endoscopy group will undergo endoscopy in 48 hours with possible stent insertion. In the ESWL group, if pain continues or aggravates, endoscopic drainage of the MPD will be carried out.

Follow-up will consists of telephone interview1 after treatment and clinical examination every 6 months thereafter. Data collected will include clinical presentation, ESWL, endoscopic and surgical procedures, life quality. In addition, S-MRCP will be performed 6 months after treatment. Blood glucose, insulin, stool elastase will be taken each clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* painful chronic pancreatitis(abdominal pain attack during the preceding 12 months);
* at least 1 calcified stone greater than 5 mm in one of its axes in the cephalic or corporeal portion of the main pancreatic duct with upstream duct dilation;
* no ERCP or ESWL carried out before admission

Exclusion Criteria:

* suspected to have malignant tumors;
* history of pancreatic surgery or gastrojejunostomy (Billroth II);
* pancreatic collection greater than 2 cm in diameter at magnetic resonance or CT scan;
* age below 18 years;
* pregnancy or lactation;
* refuse to write informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain score as accessed by izbichi pain score at 12 month | 12 months
  Whether pain is relieved depends on the change of Izbicki pain score at the baseline and 12 months after the procedure(ERCP alone or ERCP combined with ERCP). Izbicki pain score is composed of 4 parts, that is frequency of pain attacks(daily counts for 100, several times a week counts for 75, several times a month counts for 50, several times a year counts for 25 and several times a year counts for 0), VAS(subjective evaluation of pain by patients from no pain which is 0 points to imaginative maximum of pain which is 100 points), analgesic medication(morphine consumption is 100, buprenorphine is 80, pethidine is 20, tramaldol is 15, metamizole is 3 and acetylsalicylacid is 1) and time of disease-related inability to work(permanet is 100, ≤1 month is 50, ≤1 week is 25 and no inability to work during the last year is 0). Each part counts for 100 points in all.

SECONDARY OUTCOMES:
exocrine function of the pancreas through determination of fecal elastase as assessed by fecal elastase kit | 12 months
  Pancreatic exocrine function insufficiency(PEI) is defined as fecal elastase <200 μg/g. The result wii be divided into 4 conditions, that is exocrine function normal, PEI develop, PEI resolve, PEI persist.
clearance of pancreatic stones | 12 months
  Clearance of pancreatic stone is regarded as complete when clearance rate is more than 90%, partial is regarded as 50% to 90%, the rest is unsuccessful.
decompression rate of the pancreatic duct as the change of pancreatic duct diameter assessed by S-MRCP | 12 months

OTHER OUTCOMES:
complication rate | 1 months
  Complications involve pancreatitis, hemorrhage, perforation, infection and steinstrasse.
endocrine function as assessed by the combination of fasting blood glucose, insulin, C peptide, glycosylated hemoglobin | 12 months
  As mentioned earlier, the result of pancreatic endocrine function can also be divided into 4 parts similar to that of pancreatic exocrine function.
treatment-related cost from initial treatment to the end of the study(12 months) | 12 months
life quality as assessed by SF-36 questionnaire | 12 months
BMI in kg/m^2 | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No